CLINICAL TRIAL: NCT02274311
Title: Clomiphene Citrate for Treatment of Acromegaly Not Controlled by Conventional Therapies
Brief Title: Clomiphene Citrate for Treatment of Acromegaly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Felipe Henning Gaia Duarte (Other)
Responsible Party: Sponsor-Investigator, Felipe Henning Gaia Duarte, MD, PhD, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ClomipheneAcro
Record Dates: First submitted 2014-10-20; First posted 2014-10-24 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Acromegaly
Keywords: Acromegaly; SERM; Clomiphene
MeSH Terms: conditions — Acromegaly | interventions — Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clomiphene citrate (Experimental): Patients receiving clomiphene citrate
  Interventions: Drug: Clomiphene Citrate

INTERVENTIONS:
Drug: Clomiphene Citrate — Clomiphene citrate, 50 mg, orally for three months
  Other Names: Clomid; Serophene; Indux

SUMMARY:
To assess the impact of clomiphene citrate on serum insulin like growth factor 1 and testosterone levels in male acromegalic patients not controlled by surgery, radiotherapy and/or medical treatments (somatostatin analogues, dopamine agonists and/or growth hormone receptor antagonist)

DETAILED DESCRIPTION:
Acromegaly, a disease caused by a growth hormone secreting pituitary adenoma, results in reduced life span. Despite the many modalities available to treat this disease,as surgery, medical treatment and radiotherapy, uncontrolled disease persists in a significant portion of patients

Oral estrogens, alone or in combination with somatostatin receptor analogues, have been shown to control acromegaly in women. Selective estrogen receptor modulators (SERMs) resulted in similar effects in both genders. Clomiphene citrate, a SERM that increases luteinizing hormone and follicle stimulating hormone secretion, improves hypogonadism and fertility outcomes.

The aim of this study is to assess the impact of clomiphene citrate on serum insulin like growth factor 1 and testosterone levels in male acromegalic patients not controlled by surgery, radiotherapy and/or medical treatment.

In this prospective, open label, single center trial, sixteen male patients were studied. Clomiphene citrate (50 mg/day) was added to previous medical treatment for 3 months and hormonal assessment was performed prior to and during the intervention. Hormones included: growth hormone, insulin like growth factor, total testosterone, follicle stimulating hormone, luteinizing hormone and prostate-specific antigen.

ELIGIBILITY:
Inclusion Criteria:

* patients with active acromegaly on regular use of a stable dose of Octreotide-LAR and/or cabergoline for at least one year,
* Insulin like growth factor 1 above the reference range during the last year of follow-up and
* testosterone levels within or below the third inferior tertile of normality.

Exclusion Criteria:

* radiotherapy in the last 10 years, previous venous embolism (including family members),
* previous prostatic cancer or symptomatic benign hypertrophy,
* triglyceride levels above 400 mg/dL,
* renal failure defined by estimative of renal filtration below 30 ml/min,
* liver disease defined by hepatic enzymes 3 times above normal limit,
* active oncologic disease in the last 10 years and previous cardiac or cerebrovascular disease.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcello D Bronstein, MD, PhD, Study Chair — Unit of Neuroendocrinology, Discipline of Endocrinology, Department of Internal Medicine Clinical Hospital of the University of São Paulo Medical School, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Acromegalic patients with uncontrolled hormonal levels despite current medical treatment
Pre-assignment Details: Patients should be on stable medical treatment for at least 6 months prior entering the study. Patients submitted to radiotherapy in the last 10 years were not eligible.
Groups:
- Clomiphene Citrate: Patients receiving clomiphene citrate
  Clomiphene Citrate: Clomiphene citrate, 50 mg, orally for three months
  16 patients were enrolled
Period: Three Months of Clomiphene Treatment
Arm/Group | Clomiphene Citrate
Started | 16
Completed | 16
Not Completed | 0
Period: Three Months of Clomiphene Wash-out
Arm/Group | Clomiphene Citrate
Started | 16
Completed | 15
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Clomiphene Citrate: Patients receiving clomiphene citrate Clomiphene Citrate: Clomiphene citrate, 50 mg, orally for three months
  Patients with active acromegaly, defined by high IGF-1 levels, on regular use of a stable dose of Octreotide-LAR and/or Cabergoline for at least 1 year; IGF-1 above the reference range during the last year of follow-up; and T levels within or below the third inferior tertile of normality.
Arm/Group | Clomiphene Citrate
Number analyzed (Participants) | 16
Age, Customized [Median (Full Range); unit: years] | 52.5 [36 to 79]
Sex: Female, Male [Count of Participants; unit: Participants] — Only male patients were recruited
  Participants
    Female | 0
    Male | 16

OUTCOME MEASURES:

1. Primary Outcome: IGF-1 Levels
Description: The objective is to compare the change of IGF-1 value assessed in the beginning of the study (day 0), with the value obtained after three months of use of clomiphene citrate (day 90).
Time Frame: Day 90
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Clomiphene Citrate: Patients receiving clomiphene citrate
  Clomiphene Citrate: Clomiphene citrate, 50 mg, orally for three months
  16 patients were enrolled.
  IGF-1 values were assessed at D0 (baseline) and D90 (mean values)
Arm/Group | Clomiphene Citrate
Number analyzed (Participants) | 16
ng/mL | 424 (108)
Statistical Analysis 1: Comparison: Clomiphene Citrate; Measures of central tendency (mean) and variability (range and/or SD) were used to describe numeric variables. Paired Student's t test was used to verify the mean differences between dependent normally distributed variables. Wilcoxon sign test was performed to non-normally distributed dependent variables. Asignificance level of 5%was adopted for all statistical tests (P <.05); Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Testosterone Levels
Description: The objective is to compare the change of testosterone value assessed in the beginning of the study (day 0), with the value obtained after three months of use of clomiphene citrate (day 90).
Time Frame: D90
Population: 10 acromegalic patients were assessed, the other 6 patients did not have testosterone levels assessed.
Measure: Median (Standard Deviation); unit: ng/dL
Arm/Group | Clomiphene Citrate
Number analyzed (Participants) | 10
ng/dL | 282 (210)

3. Secondary Outcome: PSA Levels
Description: The objective is to compare the change of PSA value assessed in the beginning of the study (day 0), with the value obtained after three months of use of clomiphene citrate (day 90).
Time Frame: Day 90
Measure: Median (Standard Deviation); unit: ng/mL
Arm/Group | Clomiphene Citrate
Number analyzed (Participants) | 16
ng/mL | 2.0 (2.0)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at D90 (3 months after the begging of the study)
Groups:
- Clomiphene Citrate: Patients receiving clomiphene citrate
  Clomiphene Citrate: Clomiphene citrate, 50 mg, orally for three months
  No adverse events were reported
Arm/Group | Clomiphene Citrate
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No